CLINICAL TRIAL: NCT00577460
Title: Long-term Safety Study of Open-label Pramipexole Extended Release (ER) in Patients With Advanced Parkinson's Disease (PD)
Brief Title: Long-term Safety Study of Open-label Pramipexole ER in Patients With Advanced PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 248.634; 2007-004235-37 (EudraCT Number: EudraCT)
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Results first posted 2011-07-14 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

ARMS (2):
- Pramipexole (Active Comparator): Patients to receive Pramipexole ER 0.375 - 4.5 mg in tablet form daily
  Interventions: Drug: Pramipexole
- Placebo (Placebo Comparator): Patients to receive placebo tablets identical to Pramipexole ER tablets only during transfer phase
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pramipexole — Pramipexole ER 0.375 -4.5 mg
  Arms: Pramipexole
Drug: Placebo — Placebo tablets identical to Pramipexole ER tablets
  Arms: Placebo

SUMMARY:
The general aim of this study is to obtain long-term safety and tolerability data on pramipexole extended release (ER), in daily doses from 0.375mg to 4.5mg once daily (qd), in patients who have previously completed a pramipexole double-blind study in advanced Parkinson's disease (PD) (248.525 trial).

ELIGIBILITY:
Inclusion criteria:

1. Completion of the double-blind trial 248.525
2. Male or female patient with advanced idiopathic Parkinson's disease (PD), with a Modified Hoehn and Yahr stage of 2 to 4 at on-time, and a concomitant treatment with standard or controlled release L-Dopa+, or a combination of L-Dopa+ and entacapone.
3. Patient willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures. In particular the patient should be able to recognise the off-time and on-time periods during waking hours and the patient (or a family member or a guardian) should be able to record them accurately in the patient diary.
4. Signed informed consent obtained before any study procedures are carried out (in accordance with International Conference of Harmonization - Good Clinical Practice (ICH-GCP) guidelines and local legislation).

Exclusion criteria:

1. Patients prematurely withdrawn from the double-blind trial 248.525
2. Atypical parkinsonian syndromes due to drugs, metabolic disorders, encephalitis or degenerative diseases
3. Any psychiatric disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV criteria that could prevent compliance or completion of the study and/or put the patient at risk if he/she takes part in the study
4. History of psychosis, except history of drug induced hallucinations
5. History of deep brain stimulation
6. Clinically significant ECG abnormalities at baseline
7. Clinically significant hypotension and/or symptomatic orthostatic hypotension at baseline
8. Malignant melanoma or history of previously treated malignant melanoma
9. Any other clinically significant disease, whether treated or not, that could put the patient at risk or could prevent compliance or completion of the study
10. Pregnancy or breast-feeding
11. Sexually active female of childbearing potential not using a medically approved method of birth control
12. Serum levels of aspartate transaminase (AST) (serum glutamic oxaloacetic transaminase (SGOT)), alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase) (SGPT)), alkaline phosphatase (AP) or bilirubin > 2 upper limit normal (ULN) at baseline
13. Patients with a creatinine clearance < 50 mL/min at baseline
14. Any medication with central dopaminergic antagonist activity within 4 weeks prior to the baseline visit
15. Any of the following drugs within 4 weeks prior to baseline visit: methylphenidate, cinnarizine, amphetamines
16. Flunarizine within 3 months prior to baseline
17. Known hypersensitivity to pramipexole or its excipients
18. Drug abuse, according to investigators judgement, within 2 years prior to baseline
19. Participation in investigational drug studies other than the trial 248.525, or use of other investigational drugs within one month or five times the half-life of the investigational drug (whichever is longer) prior to baseline

Min Age: 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2007-12; Primary Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (70):
- 248.634.43005 Boehringer Ingelheim Investigational Site, Linz, Austria
- Czechia (5):
  - 248.634.42003 Boehringer Ingelheim Investigational Site, Pardubice
  - 248.634.42001 Boehringer Ingelheim Investigational Site, Prague
  - 248.634.42005 Boehringer Ingelheim Investigational Site, Rakovník
  - 248.634.42002 Boehringer Ingelheim Investigational Site, Rychnov nad Kněžnou
  - 248.634.42004 Boehringer Ingelheim Investigational Site, Valašské Meziříčí
- Hungary (4):
  - 248.634.36005 Boehringer Ingelheim Investigational Site, Győr
  - 248.634.36003 Boehringer Ingelheim Investigational Site, Kecskemét
  - 248.634.36006 Boehringer Ingelheim Investigational Site, Szeged
  - 248.634.36004 Boehringer Ingelheim Investigational Site, Veszprém
- India (6):
  - 248.634.91002 Boehringer Ingelheim Investigational Site, Chennai
  - 248.634.91001 Boehringer Ingelheim Investigational Site, Delhi
  - 248.634.91003 Boehringer Ingelheim Investigational Site, Hyderabad
  - 248.634.91007 Boehringer Ingelheim Investigational Site, Indore
  - 248.634.91005 Boehringer Ingelheim Investigational Site, Karnataka
  - 248.634.91006 Boehringer Ingelheim Investigational Site, Pune
- Italy (8):
  - 248.634.39001 Boehringer Ingelheim Investigational Site, Catania
  - 248.634.39010 Boehringer Ingelheim Investigational Site, Catanzaro
  - 248.634.39009 Boehringer Ingelheim Investigational Site, Chieti
  - 248.634.39007 Boehringer Ingelheim Investigational Site, Grosseto
  - 248.634.39002 Boehringer Ingelheim Investigational Site, Napolii
  - 248.634.39008 Boehringer Ingelheim Investigational Site, Pisa
  - 248.634.39005 Boehringer Ingelheim Investigational Site, Roma
  - 248.634.39011 Boehringer Ingelheim Investigational Site, Roma
- Philippines (8):
  - 248.634.63202 Boehringer Ingelheim Investigational Site, Cruz, Manila
  - 248.634.63207 Boehringer Ingelheim Investigational Site, Ermita, Manila
  - 248.634.63210 Boehringer Ingelheim Investigational Site, Makati City
  - 248.634.63205 Boehringer Ingelheim Investigational Site, Manila
  - 248.634.63206 Boehringer Ingelheim Investigational Site, Manila
  - 248.634.63201 Boehringer Ingelheim Investigational Site, Pasig
  - 248.634.63208 Boehringer Ingelheim Investigational Site, Quezon
  - 248.634.63204 Boehringer Ingelheim Investigational Site, Quezon City
- Poland (3):
  - 248.634.48001 Boehringer Ingelheim Investigational Site, Gdansk
  - 248.634.48003 Boehringer Ingelheim Investigational Site, Krakow
  - 248.634.48002 Boehringer Ingelheim Investigational Site, Warsaw
- Russia (6):
  - 248.634.07001 Boehringer Ingelheim Investigational Site, Moscow
  - 248.634.07002 Boehringer Ingelheim Investigational Site, Moscow
  - 248.634.07003 Boehringer Ingelheim Investigational Site, Moscow
  - 248.634.07004 Boehringer Ingelheim Investigational Site, Moscow
  - 248.634.07007 Boehringer Ingelheim Investigational Site, Moscow
  - 248.634.07006 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Slovakia (4):
  - 248.634.42104 Boehringer Ingelheim Investigational Site, Bratislava
  - 248.634.42105 Boehringer Ingelheim Investigational Site, Bratislava
  - 248.634.42103 Boehringer Ingelheim Investigational Site, Dubnica nad Váhom
  - 248.634.42101 Boehringer Ingelheim Investigational Site, Trnava
- South Korea (8):
  - 248.634.82001 Boehringer Ingelheim Investigational Site, Gyeonggi-do
  - 248.634.82008 Boehringer Ingelheim Investigational Site, Kyeonggi-do
  - 248.634.82007 Boehringer Ingelheim Investigational Site, Pusan
  - 248.634.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 248.634.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 248.634.82004 Boehringer Ingelheim Investigational Site, Seoul
  - 248.634.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 248.634.82006 Boehringer Ingelheim Investigational Site, Seoul
- Spain (6):
  - 248.634.34001 Boehringer Ingelheim Investigational Site, Alcorcon (Madrid)
  - 248.634.34003 Boehringer Ingelheim Investigational Site, Barcelona
  - 248.634.34004 Boehringer Ingelheim Investigational Site, Barcelona
  - 248.634.34005 Boehringer Ingelheim Investigational Site, Madrid
  - 248.634.34002 Boehringer Ingelheim Investigational Site, San Cugat Del Valles (Barcelona)
  - 248.634.34008 Boehringer Ingelheim Investigational Site, Tarrasa (Barcelona)
- Sweden (3):
  - 248.634.46005 Boehringer Ingelheim Investigational Site, Malmo
  - 248.634.46002 Boehringer Ingelheim Investigational Site, Nyköping
  - 248.634.46001 Boehringer Ingelheim Investigational Site, Stockholm
- Ukraine (6):
  - 248.634.38003 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 248.634.38006 Boehringer Ingelheim Investigational Site, Kharkiv
  - 248.634.38002 Boehringer Ingelheim Investigational Site, Kiev
  - 248.634.38004 Boehringer Ingelheim Investigational Site, Kiev
  - 248.634.38001 Boehringer Ingelheim Investigational Site, Zaporizhzhya
  - 248.634.38005 Boehringer Ingelheim Investigational Site, Zaporizhzhya
- United Kingdom (2):
  - 248.634.44007 Boehringer Ingelheim Investigational Site, Blackburn
  - 248.634.44003 Boehringer Ingelheim Investigational Site, Salford

RESULTS

PARTICIPANT FLOW:
Groups:
- PPX ER (Previous Placebo): Pramipexole ER Treatment with placebo in previous trial
- PPX ER (Previous PPX ER): Pramipexole ER Treatment with Pramipexole ER in previous trial
- PPX ER (Previous PPX IR): Pramipexole ER Treatment with Pramipexole Immediate Release (IR) in previous trial
Period: Overall Study
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Started | 129 | 123 | 139
Completed | 113 | 104 | 112
Not Completed | 16 | 19 | 27
Not completed — Adverse Event | 11 | 7 | 14
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 3 | 4
Not completed — Withdrawal by Subject | 5 | 5 | 6
Not completed — Other | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Treated Set, all patients dispensed study drug and documented to have taken at least one dose
Groups:
- PPX ER (Previous PPX IR): Pramipexole ER Treatment with Pramipexole IR in previous trial
- Total: Total of all reporting groups
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR) | Total
Number analyzed (Participants) | 129 | 123 | 139 | 391
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (9.7) | 61.7 (9.8) | 61.8 (9.7) | 61.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 55 | 65 | 178
  Male | 71 | 68 | 74 | 213

OUTCOME MEASURES:

1. Secondary Outcome: Patients Successfully Switched From Pramipexole (PPX) IR or ER to ER Assessed on UPDRS II+III
Description: Unified Parkinson's Disease Rating Scale (UPDRS) Successfully switched means: UPDRS II+III baseline score >20 without a relative worsening of UPDRS II+III score > 15% from baseline or UPDRS II+III baseline score <=20 without an absolute worsening of UPDRS II+III score > 3 from baseline UPDRS II+III ranging from 0 (normal) to 160 (severe). UPDRS part II measures activities of daily living, part III measures motor symptoms
Time Frame: One week
Population: Patients from Full Analysis Set (FAS included all patients who were dispensed study medication, had received at least one dose of study drug and had provided any post-baseline efficacy assessment) and who maintain the final dose of the previous study
Measure: Number; unit: Patients
Arm/Group | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 105 | 123
Patients | 88 | 106

2. Secondary Outcome: UPDRS II+III Change From Open Label (OL) Baseline
Description: UPDRS II+III ranging from 0 (normal) to 160 (severe). UPDRS part II measures activities of daily living, part III measures motor symptoms
Time Frame: OL Baseline and week 80
Population: Patients from FAS with values of UPDRS II+III at week 80
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 113 | 102 | 112
Scores on a scale | -3.6 (1.5) | 1.1 (1.6) | 2.5 (1.5)
Statistical Analysis 1: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX ER); PPX ER versus Placebo; Test type: Superiority or Other; p = 0.0039, ANCOVA; Analysis of covariance (ANCOVA) with factors treatment and country and covariate OL baseline
Statistical Analysis 2: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX IR); PPX IR versus Placebo; Test type: Superiority or Other; p = 0.0001, ANCOVA; Analysis of covariance (ANCOVA) with factors treatment and country and covariate OL baseline

3. Secondary Outcome: Number of Participants With UPDRS II+III Response
Description: A response means an improvement of >=20% in UPDRS II+III from OL baseline UPDRS II+III ranging from 0 (normal) to 160 (severe). UPDRS part II measures activities of daily living, part III measures motor symptoms
Time Frame: Week 80
Population: Patients from FAS with values of UPDRS II+III at week 80
Measure: Number; unit: Patients
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 113 | 102 | 112
Patients | 35 | 30 | 31

4. Secondary Outcome: Number of Patients Successfully Switched From PPX IR or ER to ER Assessed on Off-time
Description: A patient was considered as successfully switched if he/she has converted to ER without a worsening of off time by more than 12.5% from baseline. Off-time is based on patient diary data and describes a period when the patient experiences increased parkinsonian symptoms (e.g. immobility or inability to move with ease).
Time Frame: One week
Population: Patients from FAS and who maintain the final dose of the previous study
Measure: Number; unit: Patients
Arm/Group | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 95 | 110
Patients | 57 | 70

5. Secondary Outcome: Percentage Off Time During Waking Hours Total Score: Change From Baseline
Description: Percentage off-time based on patient diary data, percentage ranging from 0 (best case) to 100 (worst case). Off-time describes a period when the patient experiences increased parkinsonian symptoms (e.g. immobility or inability to move with ease).
  A negative change implies improvement
Time Frame: Baseline and week 80
Population: Patients from FAS with values of UPDRS II+III at week 80
Measure: Least Squares Mean (Standard Error); unit: percentage during waking hours
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 108 | 100 | 108
percentage during waking hours | -1.5 (2.0) | -0.3 (2.1) | 1.7 (2.0)
Statistical Analysis 1: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX ER); Test type: Superiority or Other; p = 0.5590, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate
Statistical Analysis 2: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX IR); Test type: Superiority or Other; p = 0.1289, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate

6. Secondary Outcome: Number of Participants With Response in Percentage Off Time During Waking Hours
Description: Response means >=20% improvement relative to OL baseline in the % off-time during waking hours
Time Frame: 80 weeks
Population: Patients from FAS with values of off time during waking hours at 80 weeks
Measure: Number; unit: Patients
Groups:
- Total PPX ER: Pramipexole ER, all patients
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR) | Total PPX ER
Number analyzed (Participants) | 97 | 91 | 94 | 282
Patients | 35 | 40 | 28 | 103

7. Secondary Outcome: Percentage on Time Without Dyskinesia During Waking Hours: Change From Baseline After 80 Weeks
Description: Percentage on-time based on patient diary data, percentage ranging from 0 (worst case) to 100 (best case). On-time describes a period when the patient has no symptoms of off-time and is not asleep. A positive change implies improvement.
Time Frame: Baseline and week 80
Population: Patients from FAS with values of on time during waking hours at week 80
Measure: Least Squares Mean (Standard Error); unit: percentage during waking hours
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 108 | 100 | 108
percentage during waking hours | -1.6 (2.5) | 2.9 (2.7) | -2.0 (2.6)
Statistical Analysis 1: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX ER); Test type: Superiority or Other; p = 0.1073, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate
Statistical Analysis 2: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX IR); Test type: Superiority or Other; p = 0.8694, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate

8. Secondary Outcome: Percentage on Time With Non Troublesome Dyskinesia During Waking Hours: Change From Baseline After 80 Weeks
Description: Percentage on-time with non troublesome dyskinesia based on patient diary data, percentage ranging from 0 (worst case) to 100 (best case). On-time describes a period when the patient has no symptoms of off-time and is not asleep. A positive change implies improvement
Time Frame: Baseline and week 80
Population: Patients from FAS with values of on time during waking hours at week 80
Measure: Least Squares Mean (Standard Error); unit: percentage during waking hours
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 108 | 100 | 108
percentage during waking hours | 3.8 (1.8) | -2.7 (1.9) | 0.2 (1.8)
Statistical Analysis 1: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX ER); Test type: Superiority or Other; p = 0.0009, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate
Statistical Analysis 2: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX IR); Test type: Superiority or Other; p = 0.0573, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate

9. Secondary Outcome: Percentage on Time Without Dyskinesia or With Non Troublesome Dyskinesia During Waking Hours: Change From Baseline After 80 Weeks
Description: Percentage on-time without dyskinesia or with non troublesome dyskinesia based on patient diary data, percentage ranging from 0 (worst case) to 100 (best case). On-time describes a period when the patient has no symptoms of off-time and is not asleep. A positive change implies improvement
Time Frame: Baseline and week 80
Population: Patients from FAS with values of on time during waking hours at week 80
Measure: Least Squares Mean (Standard Error); unit: percentage during waking hours
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 108 | 100 | 108
percentage during waking hours | 1.8 (2.2) | 0.7 (2.3) | -0.9 (2.3)
Statistical Analysis 1: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX ER); Test type: Superiority or Other; p = 0.6434, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate
Statistical Analysis 2: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX IR); Test type: Superiority or Other; p = 0.2469, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate

10. Secondary Outcome: Percentage on Time With Troublesome Dyskinesia During Waking Hours: Change From Baseline After 80 Weeks
Description: Percentage on-time with troublesome dyskinesia based on patient diary data, percentage ranging from 0 (worst case) to 100 (best case). On-time describes a period when the patient has no symptoms of off-time and is not asleep. A positive change implies improvement
Time Frame: Baseline and week 80
Population: Patients from FAS with values of on time during waking hours at week 80
Measure: Least Squares Mean (Standard Error); unit: percentage during waking hours
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 108 | 100 | 108
percentage during waking hours | -0.4 (1.0) | -0.3 (1.1) | -0.7 (1.1)
Statistical Analysis 1: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX ER); Test type: Superiority or Other; p = 0.9741, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate
Statistical Analysis 2: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX IR); Test type: Superiority or Other; p = 0.7620, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate

11. Secondary Outcome: Number of Participants With Response in CGI-I
Description: Clinical Global Impression of Improvement (CGI-I), CGI-I scores ranging from '1' (very much improved) to '7' (very much worse). For patients previously treated with Placebo, all patients with at least "much improved" were considered as responders. For patients previously treated with PPX ER or IR, all patients with no change to very much improved were considered as responders
Time Frame: 32 weeks
Population: Patients from FAS with values of CGI-I at week 32
Measure: Number; unit: Patients
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR) | Total PPX ER
Number analyzed (Participants) | 124 | 115 | 124 | 363
Patients | 50 | 106 | 114 | 270

12. Secondary Outcome: Number of Participants With Response in PGI-I
Description: Patient Global Impression of Improvement (PGI-I), PGI-I scores ranging from '1' (very much better) to '7' (very much worse). For patients previously treated with Placebo, all patients with at least "much better" were considered as responders. For patients previously treated with PPX ER or IR, all patients with no change to very much better were considered as responders
Time Frame: 32 weeks
Population: Patients from FAS with values of PGI-I at week 32
Measure: Number; unit: Patients
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR) | Total PPX ER
Number analyzed (Participants) | 124 | 115 | 124 | 363
Patients | 45 | 102 | 113 | 260

13. Secondary Outcome: Number of Participants With Response in PGI-I for Early Morning Off Symptoms
Description: Patient Global Impression of Improvement (PGI-I) for early morning off symptoms, PGI-I scores ranging from '1' (very much better) to '7' (very much worse). For patients previously treated with Placebo, all patients with at least "much better" were considered as responders. For patients previously treated with PPX ER or IR, all patients with no change to very much better were considered as responders
Time Frame: 32 weeks
Population: Patients from FAS with values of PGI-I for early morning off symptoms at week 32
Measure: Number; unit: Patients
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR) | Total PPX ER
Number analyzed (Participants) | 125 | 116 | 125 | 366
Patients | 45 | 103 | 112 | 260

14. Secondary Outcome: UPDRS I Total Score and Change From OL Baseline at Week 80
Description: UPDRS I ranging from 0 (normal) to 16 (severe). UPDRS I measures Mentation, Behavior and Mood
Time Frame: OL baseline and week 80
Population: Patients from FAS with values of UPDRS I at week 80
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 113 | 104 | 113
units on a scale | 0.1 (0.2) | 0.5 (0.2) | 0.5 (0.2)
Statistical Analysis 1: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX ER); Test type: Superiority or Other; p = 0.0831, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate
Statistical Analysis 2: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX IR); Test type: Superiority or Other; p = 0.0759, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate

15. Secondary Outcome: UPDRS II Total Score and Change From OL Baseline at Week 80
Description: UPDRS II ranging from 0 (normal) to 52 (severe). UPDRS Part II is calculated as the average of UPDRS part II at on and UPDRS part II at off-period for each of the 13 activities
Time Frame: OL baseline and week 80
Population: Patients from FAS with values of UPDRS II at week 80
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 113 | 102 | 112
units on a scale | -0.4 (0.5) | 0.4 (0.6) | 1.0 (0.5)
Statistical Analysis 1: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX ER); Test type: Superiority or Other; p = 0.1713, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate
Statistical Analysis 2: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX IR); Test type: Superiority or Other; p = 0.0130, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate

16. Secondary Outcome: UPDRS III Total Score and Change From OL Baseline at Week 80
Description: UPDRS III ranging from 0 (normal) to 108 (severe). UPDRS part III measures motor symptoms
Time Frame: OL baseline and week 80
Population: Patients from FAS with values of UPDRS III at week 80
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 113 | 104 | 113
units on a scale | -3.1 (1.1) | 0.7 (1.1) | 1.3 (1.1)
Statistical Analysis 1: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX ER); Test type: Superiority or Other; p = 0.0015, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate
Statistical Analysis 2: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX IR); Test type: Superiority or Other; p = 0.0002, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate

17. Secondary Outcome: UPDRS IV Total Score and Change From OL Baseline at Week 80
Description: UPDRS IV ranging from 0 (normal) to 23 (severe). UPDRS IV measures complications of therapy
Time Frame: OL baseline and week 80
Population: Patients from FAS with values of UPDRS IV at week 80
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 113 | 104 | 113
Unit on a scale | 0.0 (0.2) | -0.0 (0.3) | 0.2 (0.2)
Statistical Analysis 1: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX ER); Test type: Superiority or Other; p = 0.8760, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate
Statistical Analysis 2: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX IR); Test type: Superiority or Other; p = 0.5113, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate

18. Secondary Outcome: Parkinson Fatigue Scale (PFS-16) Score and Change From OL Baseline at Week 80
Description: PFS-16 (Parkinson fatigue scale) ranging from 16 (better perceived health status) to 80 (severe symptoms of the disease) measuring aspects of fatigue that are relevant to patients with PD
Time Frame: OL baseline and week 80
Population: Patients from FAS with values of PFS-16 score at week 80
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 116 | 106 | 114
Unit on a scale | -0.3 (1.5) | 3.8 (1.6) | 3.5 (1.6)
Statistical Analysis 1: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX ER); Test type: Superiority or Other; p = 0.0148, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate
Statistical Analysis 2: Comparison: PPX ER (Previous Placebo) vs PPX ER (Previous PPX IR); Test type: Superiority or Other; p = 0.0201, ANCOVA; Analysis of covariance with factors for treatment, country and baseline as a covariate

19. Secondary Outcome: Number of Participants With L-dopa Daily Dose Change: Change From OL Baseline at Week 80
Time Frame: OL baseline and week 80
Population: Patients from FAS with documentation of levodopa (L-DOPA) daily dose at week 80
Measure: Number; unit: Patients
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR) | Total PPX ER
Number analyzed (Participants) | 125 | 114 | 132 | 371
Patients
  Decrease | 24 | 12 | 12 | 48
  Increase | 8 | 18 | 27 | 53
  No change | 93 | 84 | 93 | 270

20. Secondary Outcome: Number of Participants With Changes in Pramipexole Doses After 80 Weeks Compared to Pramipexole Dose at OL Baseline
Time Frame: OL baseline and week 80
Population: Patients from Treated Set (all patients who were dispensed study drug and were documented to have at least one dose of investigational treatment) and treated until week 80
Measure: Number; unit: Patients
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR) | Total PPX ER
Number analyzed (Participants) | 125 | 115 | 126 | 366
Patients
  Reduced | 56 | 33 | 26 | 115
  Unchanged | 40 | 43 | 53 | 136
  Increased | 29 | 39 | 47 | 115

21. Secondary Outcome: Number of Participants With Serious Adverse Events
Time Frame: 80 weeks
Population: The Treated Set (TS) included all patients who were dispensed study drug and were documented to have at least one dose of investigational treatment
Measure: Number; unit: Patients
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR) | Total PPX ER
Number analyzed (Participants) | 129 | 123 | 139 | 391
Patients | 14 | 11 | 14 | 39

22. Primary Outcome: Percentage of Patients With Adverse Events, Adverse Drug Reactions, Serious Adverse Events
Description: The aim of this study was to obtain long-term safety and tolerability data on pramipexole ER, in patients who have previously completed a pramipexole double blind study in advanced Parkinson's Disease (PD) (248.525 (NCT00466167)). Therefore these items were considered as a safety evaluation.
Time Frame: 80 weeks
Population: Patients from Treated Set (defined as all patients who were dispensed study drug and were documented to have at least one dose of investigational treatment)
Measure: Number; unit: Percentage of participants
Groups:
- Placebo: Treatment with matching placebo in previous trial (NCT00466167)
- PPX ER: Treatment with Pramipexole ER in previous trial
- PPX IR: Treatment with Pramipexole IR in previous trial
Arm/Group | Placebo | PPX ER | PPX IR
Number analyzed (Participants) | 129 | 123 | 139
Percentage of participants
  Percentage of Patients with Adverse Events | 85.3 | 83.7 | 79.9
  Percentage of Patients with Adverse Drug Reactions | 52.7 | 48.8 | 45.3
  Percentage of Patients with Serious Adverse Events | 10.9 | 8.9 | 10.1

23. Secondary Outcome: Supine Diastolic Blood Pressure, Baseline and Week 80, Vital Signs Treated Set
Time Frame: OL Baseline and Week 80
Population: Vital Signs Treated Set - All participants treated with study drug and have both baseline and week 80 vital sign data
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 125 | 114 | 132
mm Hg
  OL Baseline | 77.4 (8.9) | 77.3 (8.6) | 77.6 (9.4)
  End of OL | 77.4 (8.9) | 78.3 (8.9) | 77.2 (8.3)

24. Secondary Outcome: Standing Diastolic Blood Pressure, Baseline and Week 80, Vital Signs Treated Set
Time Frame: OL Baseline and Week 80
Population: Vital Signs Treated Set - All participants treated with study drug and have both baseline and week 80 vital sign data
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 125 | 113 | 131
mm Hg
  OL Baseline | 77.8 (9.2) | 77.3 (9.1) | 77.6 (9.9)
  End of OL | 77.6 (9.1) | 78.1 (9.3) | 76.4 (9.7)

25. Secondary Outcome: Supine Systolic Blood Pressure, Baseline and Week 80, Vital Signs Treated Set
Time Frame: OL Baseline and Week 80
Population: Vital Signs Treated Set - All participants treated with study drug and have both baseline and week 80 vital sign data
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 125 | 114 | 132
mm Hg
  OL Baseline | 121.6 (12.2) | 124.5 (15.4) | 125.7 (14.8)
  End of OL | 124.2 (13.5) | 123.8 (14.2) | 124.4 (14.7)

26. Secondary Outcome: Standing Systolic Blood Pressure, Baseline and Week 80, Vital Signs Treated Set
Time Frame: OL Baseline and Week 80
Population: Vital Signs Treated Set - All participants treated with study drug and have both baseline and week 80 vital sign data
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 125 | 113 | 131
mm Hg
  OL Baseline | 120.2 (13.9) | 121.1 (16.4) | 120.9 (15.9)
  End of OL | 121.9 (15.0) | 121.6 (14.3) | 120.5 (16.0)

27. Secondary Outcome: Supine Pulse Rate, Baseline and Week 80, Vital Signs Treated Set
Time Frame: OL Baseline and Week 80
Population: Vital Signs Treated Set - All participants treated with study drug and have both baseline and week 80 vital sign data
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 125 | 114 | 132
beats per minute
  OL Baseline | 73.6 (9.6) | 72.6 (9.2) | 73.2 (9.0)
  End of OL | 75.8 (9.0) | 74.2 (7.9) | 74.4 (10.0)

28. Secondary Outcome: Standing Pulse Rate, Baseline and Week 80, Vital Signs Treated Set
Time Frame: OL Baseline and Week 80
Population: Vital Signs Treated Set - All participants treated with study drug and have both baseline and week 80 vital sign data
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 125 | 113 | 131
beats per minute
  OL Baseline | 78.3 (10.7) | 78.0 (9.5) | 77.7 (9.9)
  End of OL | 79.3 (8.7) | 77.7 (7.5) | 78.8 (10.4)

29. Secondary Outcome: Body Weight of Female Patients, Baseline and Week 80, Vital Signs Treated Set
Time Frame: OL Baseline and Week 80
Population: Vital Signs Treated Set - All participants treated with study drug and have both baseline and week 80 vital sign data
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 55 | 52 | 62
kg
  OL Baseline | 61.9 (13.0) | 61.7 (14.0) | 63.8 (14.6)
  End of OL | 63.6 (13.8) | 61.7 (15.0) | 63.6 (16.0)

30. Secondary Outcome: Body Weight of Male Patients, Baseline and Week 80, Vital Signs Treated Set
Time Frame: OL Baseline and Week 80
Population: Vital Signs Treated Set - All participants treated with study drug and have both baseline and week 80 vital sign data
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 70 | 62 | 70
kg
  OL Baseline | 73.0 (15.7) | 72.1 (12.2) | 70.8 (13.2)
  End of OL | 73.9 (16.4) | 72.7 (12.5) | 72.0 (14.0)

31. Secondary Outcome: Epworth Sleepiness Scale (ESS), Baseline and End of Open Label, Treated Set
Description: ESS Total score ranges from zero (best) to 24 (worst); scale has 8 items, each rated from zero (no chance of dozing) to 3 (high chance of dozing)
Time Frame: OL Baseline and Week 80
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 125 | 113 | 130
units on a scale
  OL Baseline | 7.2 (4.6) | 8.1 (4.1) | 8.1 (4.9)
  Change from baseline at end of OL | 0.5 (5.1) | 1.2 (4.7) | 1.2 (4.8)

32. Secondary Outcome: Modified Minnesota Impulsive Disorder Interview (mMIDI), Frequency of Patients With at Least One Abnormal Behavior, Treated Set
Description: The mMIDI is a semi-structured interview designed to assess impulsive control disorders. The scale was modified to focus behaviors of: pathological gambling, compulsive buying and compulsive sexual behavioral.
Time Frame: Baseline, 80 weeks
Population: Treated Set - all patients dispensed drug and documented to have taken at least one dose
Measure: Number; unit: participants
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR)
Number analyzed (Participants) | 129 | 123 | 139
participants
  Abnormal behavior - pathological gambling | 0 | 0 | 0
  Abnormal behavior - compulsive buying | 2 | 0 | 2
  Abnormal behavior - compulsive sexual behavior | 2 | 2 | 0

ADVERSE EVENTS:
Time Frame: 80 weeks
Arm/Group | PPX ER (Previous Placebo) | PPX ER (Previous PPX ER) | PPX ER (Previous PPX IR) | Total PPX ER
Serious Adverse Events (participants affected / at risk) | 14/129 | 11/123 | 14/139 | 39/391
Other Adverse Events (participants affected / at risk) | 87/129 | 74/123 | 81/139 | 242/391
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PPX ER (Previous Placebo) (N=129) | PPX ER (Previous PPX ER) (N=123) | PPX ER (Previous PPX IR) (N=139) | Total PPX ER (N=391)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 1 | 2
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Rectal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 1 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 3
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Eyeball rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Cerebellar haematoma (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Dyskinesia (Nervous system disorders) | 0 | 1 | 0 | 1
Dystonia (Nervous system disorders) | 0 | 1 | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1
On and off phenomenon (Nervous system disorders) | 0 | 0 | 1 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0 | 1
Cardiac neurosis (Psychiatric disorders) | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 1
Paramnesia (Psychiatric disorders) | 0 | 1 | 0 | 1
Pathological gambling (Psychiatric disorders) | 0 | 0 | 1 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PPX ER (Previous Placebo) (N=129) | PPX ER (Previous PPX ER) (N=123) | PPX ER (Previous PPX IR) (N=139) | Total PPX ER (N=391)
Cataract (Eye disorders) | 9 | 8 | 6 | 23
Constipation (Gastrointestinal disorders) | 8 | 5 | 3 | 16
Nausea (Gastrointestinal disorders) | 10 | 7 | 7 | 24
Nasopharyngitis (Infections and infestations) | 3 | 4 | 8 | 15
Fall (Injury, poisoning and procedural complications) | 8 | 9 | 6 | 23
Decreased appetite (Metabolism and nutrition disorders) | 4 | 5 | 8 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6 | 6 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 7 | 5 | 19
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 9 | 12
Dizziness (Nervous system disorders) | 13 | 11 | 4 | 28
Dyskinesia (Nervous system disorders) | 41 | 33 | 32 | 106
Dystonia (Nervous system disorders) | 4 | 8 | 7 | 19
Headache (Nervous system disorders) | 6 | 5 | 8 | 19
Somnolence (Nervous system disorders) | 15 | 18 | 19 | 52
Tremor (Nervous system disorders) | 6 | 4 | 8 | 18
Hallucination (Psychiatric disorders) | 10 | 6 | 6 | 22
Insomnia (Psychiatric disorders) | 10 | 10 | 7 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.